CLINICAL TRIAL: NCT02228772
Title: Phase I Study of MLN 9708 in Addition to Chemotherapy for the Treatment of Acute Lymphoblastic Leukemia in Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Philip C. Amrein, M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-200
Record Dates: First submitted 2014-08-23; First posted 2014-08-29 (Estimated); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Acute Lymphoblastic Leukemia; Lymphoblastic Lymphoma; B-cell Adult Acute Lymphoblastic Leukemia; T-cell Adult Acute Lymphoblastic Leukemia
Keywords: Acute lymphoblastic Leukemia; Lymphoblastic lymphoma; B-cell Adult Acute Lymphoblastic Leukemia; T-cell Adult Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — ixazomib; Vincristine; Cytarabine; Doxorubicin; Mercaptopurine; Cyclophosphamide; Methotrexate; merphos

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MLN 9708 (Experimental): * Dose escalation will occur using a standard 3+3 dose escalation approach, beginning in dose level I with dose cohorts and rules for escalation and de-escalation.
  * MLN 9708 will be given with standard multi-drug regimen for ALL . MLN 9708 will be administered on determined days during Induction therapy cycle and Consolidation cycle. If remission occurs and if eligible, the next stage with be either Stem Cell or Bone Marrow Transplant.
    * If not eligible to receive a transplant, the participant will continue on this study for the next 3 stages.
      * CNS Therapy
      * Consolidation 2
      * Continuation Therapy
  No further MLN9708, the investigational drug, will be given after Consolidation 1 Standard chemotherapy -Vincristine, Cytarabine, Doxorubicin, Mercaptopurine, Cyclophosphamide, Methotrexate
  Interventions: Drug: MLN 9708; Drug: Vincristine; Drug: Cytarabine; Drug: Doxorubicin; Drug: Mercaptopurine; Drug: Cyclophosphamide; Drug: Methotrexate

INTERVENTIONS:
Drug: MLN 9708 — Patients will received standard chemotherapy as well as MLN 9708 in escalating doses.
  Other Names: Ixazomib
Drug: Vincristine — Standard chemotherapy dosage and duration
  Other Names: Oncovin; Vincasar PFS; Vincrex; Vincristine sulfate; VCR
Drug: Cytarabine — Standard chemotherapy dosage and duration
  Other Names: Ara-C; Cytosar-U; Cytosine arabinoside
Drug: Doxorubicin — Standard chemotherapy dosage and duration
  Other Names: Adriamycin, Rubex
Drug: Mercaptopurine — Standard chemotherapy dosage and duration
  Other Names: 6-MP; Purinethol; Purixan
Drug: Cyclophosphamide — Standard chemotherapy dosage and duration
  Other Names: Cytoxan; Neosar; CTX
Drug: Methotrexate — Standard chemotherapy dosage and duration
  Other Names: Folex; Mexate; MTX; Methotrex (formerly Amethopterin)

SUMMARY:
This research study is evaluating a combination of drugs considered standard treatment for children and young adults with acute lymphoblastic leukemia (ALL), in combination with a new drug called MLN 9708. Additionally, the study is also evaluating if bone marrow or stem cell transplantation, which will be given to some participants, helps to prevent ALL from returning.

DETAILED DESCRIPTION:
In this research study, the investigators are studying the optimal dose of the drug MLN 9708 when given with a standard multi-drug regimen. In the first part of the study, up to 18 participants will be enrolled at different doses of MLN 9708. Once the maximally tolerated (highest, safest dose) is established, an additional 10 participants will be enrolled.

Additionally, bone marrow (tissue found in the inside of bones) or stem cell transplantation will be given to some participants to study whether it helps to prevent ALL from returning.

The study treatment consists of several different stages

* Induction
* Consolidation 1
* Or Stem Cell or Bone Marrow Transplant (if you are eligible based on your medical condition and the availability of a matched stem cell donor)
* Or If you do not have a transplant:

  * CNS Therapy
  * Consolidation 2
  * Continuation Therapy

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphoblastic leukemia, excluding known mature B-cell ALL by the presence of any of the following: surface immunoglobulin, L3 morphology, t(8;14)(q24;q32), t(8;22), or t(2;8).
* Patients with mature B-cell ALL will be removed from the protocol as soon as that diagnosis is made and should be treated on a B-cell leukemia (Burkitt's) protocol. NOTE: Patients with T-cell surface markers and a t(8;14)(q24;q11) remain eligible.
* Patients with lymphoblastic lymphoma are also eligible
* No prior anti-leukemic therapy except the following are allowed: <1 week of corticosteroids, or hydroxyurea or emergent leukopheresis. Longer steroid use for diseases other than leukemia is permitted.
* Age 51- 75 years
* Voluntary written consent must be given before performance of any study-related procedures not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
* If patient is known to be HIV positive, they will not be eligible for the protocol. HIV testing is not mandatory prior to protocol enrollment.
* Patients whose comorbid medical condition, in the investigator's opinion, would make participation in this trial and adherence to the protocol guidelines difficult should be excluded.
* Patients with an active psychiatric or mental illness making informed consent or careful clinical follow-up unlikely are excluded.
* Ejection fraction ≥ 45%
* Creatinine<2.0 times upper limit of normal
* Total bilirubin < 1.5 times upper limit of normal except for known conjugation diseases such as Gilbert's, ALT and AST <3.0 times upper limit of normal. Direct bilirubin is not an inclusion criteria.
* ECOG performance status of 0, 1, 2
* Non pregnant and non lactating Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, AND
  * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Male patients, even if surgically sterilized (i.e., status post-vasectomy), must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)

Exclusion Criteria:

* Patients meeting any of the following exclusion criteria are not to be enrolled in the study.
* Female patients who are lactating or have a positive serum pregnancy test during the screening period.
* Major surgery within 14 days before enrollment. Biopsies and line placement procedures are not exclusion criteria.
* Radiotherapy within 14 days before enrollment. Radiotherapy is excluded during induction and consolidation 1 while receiving MLN 9708.
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
* Active hepatitis B or C virus infection, or known human immunodeficiency virus (HIV) positive. Hepatitis and HIV testing are not required prior to the start of treatment.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
* Patient has ≥ Grade 3 peripheral neuropathy, or Grade 2 with pain on clinical examination during the screening period.
* Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of MLN9708 including difficulty swallowing.
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 21days of the start of this trial and throughout induction and consolidation 1 portions of this trial (while on MLN 9708). Patients may enroll in transplant and post transplant studies after consolidation 1 treatment (See Section 6.5).
* Systemic treatment, within 14 days before the first dose of MLN9708, with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort. Ciprofloxocin should not be administered for at least 2 days before MLN 9708 administration. Extended release ciprofloxocin should not be administered for at least 3 days prior to MLN 9708 administration.

Ages: 51 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Maximum Dose Tolerated of MLN 9708 | 2 Years

SECONDARY OUTCOMES:
Percentage of Patient with Complete Remission (CR) rate at the end of induction therapy | 30 Days
Percentage of Participants with Disease Free Survival | 2 Years
Rate of Overall survival (OS) | 1 Year, 2 Year, 3 Year
Complete Remission Rate | 2 Years
Rate of Toxicity | 2 Years
  Assess adverse events, serious adverse events, neurotoxicity grading

CONTACTS AND LOCATIONS:
Overall Officials: Philip Amrein, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts